CLINICAL TRIAL: NCT00383461
Title: Computerized EMR-Assisted Smoking Cessation (CEASCE)
Brief Title: Computer-Based Stop Smoking Program in Assisting Doctors in Helping Adults Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer S. Haas, MD, MSPH, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Masking: None
Other Study IDs: BWH-2004-P-001029/2; R21CA121906 (NIH)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco use disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: smoking cessation intervention
Other: counseling intervention

SUMMARY:
RATIONALE: Computer-based stop smoking programs may assist doctors in helping patients stop smoking.

PURPOSE: This randomized clinical trial is studying how well a computer-based stop smoking program works in assisting doctors in helping adults stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop an electronic medical record (EMR)-based strategy, the Computerized EMR-Assisted Smoking Cessation Effort (CEASCE), for assisting physicians in treating tobacco use in adults who are currently smokers.
* Assess the reach and effectiveness of CEASCE by conducting a randomized controlled trial in the Brigham and Women's Primary Care Practice-Based Research Network to determine its effectiveness in increasing the proportion of smokers who receive treatment.
* Assess the adoption, implementation, and short-term maintenance of CEASCE by measuring the proportion and characteristics of providers who use CEASCE, the consistency with which providers use the components of CEASCE, and changes in the use of CEASCE over time.

OUTLINE: This is a randomized, controlled, multicenter study. Clinics are stratified according to socioeconomic mix of patients and clinic type (community health center vs hospital based vs community-based). Clinics are randomized to 1 of 2 intervention arms.

* Arm I (intervention): Primary care providers utilize the Computerized Electronic Medical Record (EMR)-Assisted Smoking Cessation Effort (CEASCE) decision support system comprising a 5-step algorithm (i.e., the "5 A's"). CEASCE provides reminders to primary care providers to document smoking status using the "5 A's" (Ask, Advise, Assess, Assist, and Arrange). Primary care providers input information into the CEASCE, including asking the patient about their smoking status (Ask), the date they advised the patient to quit (Advise), an assessment of the patient's readiness to quit (Assess), and the action that was taken by the physician (Assist). When the primary care provider inputs information, CEASCE automatically presents actions that are tailored to the smoker's readiness to quit. Actions offered include setting a quit date, prescribing medications, referral to a smoking-cessation counselor, discussing barriers to quitting, counseling about the health risks of smoking, and an offer to help the smoker when she is ready to quit. CEASCE automatically prints educational materials and sends an e-mail to a smoking cessation counselor for patients who are agreeable to having a smoking cessation counselor contact them. The smoking cessation counselor makes 4 attempts to contact the patient by telephone within 30 days. If the patient is ready, the counselor facilitates enrollment into a smoking cessation program and documents the outcome of the referral. The referring primary care provider then receives an e-mail message regarding the outcome.

Primary care providers complete surveys after ≥ 6 months of experience with the intervention. Some patients participate in an exit interview immediately after their primary care visit.

* Arm II (control): Patients receive current standard of care, including documentation of smoking status and contact from a smoking-cessation counselor only after receiving a referral.

PROJECTED ACCRUAL: A total of 4,314 participants (primary care providers and patients) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Primary care providers and their patients in the Brigham and Women's Primary Care Practice-Based Research Network
* Patient is currently a smoker

PATIENT CHARACTERISTICS:

* Must speak English or Spanish
* No significant cognitive impairment (e.g., dementia or active psychosis)

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4314 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Haas, MD, MSPH, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts

REFERENCES:
- [Derived] Linder JA, Rigotti NA, Schneider LI, Kelley JH, Brawarsky P, Haas JS. An electronic health record-based intervention to improve tobacco treatment in primary care: a cluster-randomized controlled trial. Arch Intern Med. 2009 Apr 27;169(8):781-7. doi: 10.1001/archinternmed.2009.53. PMID 19398690